# Modifying and Evaluating Virtual Reality Job Interview Training for Youth in Transition

Consent to participate in a Research Study (18-26 year olds)

# **Principal Investigator:**

Matthew J. Smith, Ph.D., School of Social Work, University of Michigan

# Invitation to Participate in a Research Study

We invite you to be part of a research study to test if a new computer program improves job interviewing skills. We are asking you to be part of this study because:

- 1) You are 18-26 years old
- 2) You have a diagnosis on the autism spectrum disorder or another type of educational disability
- 3) You have an Individualized Education Plan (IEP)

# . Important Information about the Research Study

Students may have difficulty finding jobs. We created a virtual reality app to improve interviewing skills for students with a form of autism. We are asking you to be part of a research study. We want to test the virtual reality app to see if it helps improve interview skills and helps students find jobs. We plan to ask 90 students between the ages of 16 and 26 to participate in our research.

The **National Institute of Mental Health** funded this study.

# **Description of Your Involvement**

#### If you join this study:

30 students will get the usual job interview training.

60 students will get the job interview training using the virtual reality app.

Students are picked randomly (like with the flip of a coin).

## You will complete the following research visits:

#### **Before Visit 1**

You will read the consent form. This should take about 10 minutes Research staff will answer any of your questions.

You will sign the consent form if you want to join the study.

#### Visit 1 & 2

You will complete a short reading test. This should take about 10 minutes.

You will complete a baseline employment survey.

Your parent or teacher will answer some questions about your social skills.

You will complete a few learning and memory tests from the National Institute of Health toolbox IPAD application. This should take about 30 minutes.

You will complete a brief survey about your mood. This should take about 5 minutes.

You will complete one practice job interview role-play with a research staff at your school. These interviews will be audio and/or video recorded. You must agree to the video and audio recordings if you are going to participate. This should take about 25 minutes. Then you will complete 3 brief self-report surveys about your anxiety, motivation, and self-confidence. This should take about 25 minutes.

#### After Visit 2

You will be picked at random (similar to a flip of a coin) to use the virtual reality training or usual job interview training. Students chosen for the usual job training will get to use the virtual reality training after they complete the study.

If you are not in the virtual training group, you will skip Visits 3-16. You will rejoin the study at Visit17.

#### Visit 3

Students in the virtual training group will learn how to use the virtual training program. This should take about 45 minutes.

#### Visit 4

You will train with the educational content.

#### Visit 5

You will use 1 class period to learn to talk to the virtual Interviewer.

#### Visits 6-16

You will complete up to 3 virtual job interviews per visit.

#### Visit 17

All students in the study will complete one job interview role-play with research staff which will be video and/or audio-recorded. This should take about 25 minutes. You will complete another employment follow up survey. After that, you will complete 4 brief self-report surveys about your mood, anxiety, motivation, and self-confidence. This should take about 25 minutes. You will then complete a survey about how much you liked the virtual reality training. This should take about 5 minutes.

## 6-Month Follow-Up

You will complete a follow-up survey by phone or email.

# **Benefits of Participation**

Since the training was created to improve the ability to interview, you may receive some direct benefit from participating. We hope that what we find out in this study will help us to create better interview training for other students.

# **Risks and Discomforts of Participation**

There is a rare confidentiality risk that the University of Michigan computer server system could be breached. We will reduce this risk by storing your data on the server protected by passwords and a firewall. Spending 45 minutes using the app could cause fatigue or boredom. Please tell your teacher or a research staff member if you need a break. Also, we will offer you a 5-minute break between the virtual job interviews.

# Incentive to be in the study

## Payment Information:

You will receive a \$10.00 gift card if found to be ineligible after the reading test

You will receive a:

\$25.00 gift card for completing Visit 1

\$25.00 gift card for completing Visit 2

\$25.00 gift card for completing Visit 17

\$10.00 gift card for completing the 6-month follow-up interview.

Students will not be paid to use the intervention. At most, students can earn up to \$85. If you choose to no longer participate in the study, you will be paid whatever part(s) of the study you have completed. There are no costs to you.

# Confidentiality

We plan to share the results of this study with the public. We will not include any information that would identify you. We will protect your privacy by completing all research visits in a private or semi-private research room. To keep this information safe, the researchers will enter study data on a computer that is protected by a password. To protect your confidentiality, your name will not be in any written or published materials. The researchers will keep this information indefinitely for future research about virtual reality interventions.

There are some reasons why people other than the researchers may need to view your study information, but they will not need to see your name or personal information. The people work for organizations that make sure our research is done safely and properly. The organizations include the University of Michigan, government research offices, or the study sponsor, the National Institute of Mental Health.

A description of this study will be posted on a public website, <a href="http://ClincalTrials.gov">http://ClincalTrials.gov</a>, and summary results of this study will be posted on this website at the conclusion of the research, as required by the National Institutes of Health (NIH), the study sponsor. No information that can identify you will be posted.

## What will happen to the information we collect about you after the study is over?

We will store your data to use for future research studies. Your name and any other identifying information will be secured and stored separately from your research data at the School of Social Work. Only Dr. Smith, the Principal Investigator and study team members, will have access to your research files and data. Research data may be shared with other investigators but will never contain any information that could identify you. For example, the cognitive assessment data will be sent to a licensed neuropsychologist for analysis. They will also create a summary report. You may receive a copy of this summary report, and, if you would like, the summary report may also be shared with your teacher and/or educational team. You may indicate your sharing preference below.

Research data will also be entered into the NIH autism database without any information that can identify you.

You will receive a summary of the findings and a copy of the primary publication. The summary report will not include any identifying information.

There is no plan to provide you with any financial benefits from commercial products derived from the data.

# **Voluntary Nature of the Study**

Participating in this study is completely voluntary. It is completely up to you whether you want to be in the study. Even if you say yes, you may change your mind and stop at any time. You may also choose to not answer a question for any reason.

If you complete a consent form, but do not complete the study in a timely manner then you will be reminded after 2 weeks to complete the study via a phone call with an email follow-up 1 week later. Then we will remind you 5-6 times for 12 weeks. After 12 weeks of non-responsiveness then you will be identified as lost-to-follow-up and we will not contact you further. We can also have you complete your post study visit at the University Of Michigan School Of Social Work.

Lastly, if you choose not to participate, this choice will not affect your relationship with the school or teachers

# **Contact Information for the Study Team**

If you have questions about this research, including questions about scheduling or your payment for participating, you may contact **Dr. Matthew Smith** at <a href="mattjsmi@umich.edu">mattjsmi@umich.edu</a> or **(734) 764-9322**.

# Contact Information for Questions about Your Rights as a Research Participant

If you have questions about your rights as a research participant, or wish to obtain information, ask questions or discuss any concerns about this study with someone other than the researcher(s), please contact the:

University of Michigan Health Sciences and Behavioral Sciences Institutional Review Board 2800 Plymouth Road Building 520, Room 1169

Ann Arbor, MI 48109-2800

Phone: (734) 936-0933 or toll free, (866) 936-0933

Email: <u>irbhsbs@umich.edu</u>

#### **Conflict of Interest Disclosure**

Dr. Matthew Smith, the principal investigator and the person responsible for the conduct of this research study, and Dr. Rogerio Pinto, a co-investigator of the study, are inventors of the Virtual Interview Training program and have a financial interest in the program. Therefore, they have the potential, in appearance or reality, to bias the research. Our Institutional Review Board has reviewed this case and developed a conflict management plan to address the conflict of interest. Safeguards are in place to assure objectivity of the research study.

| 0- | | _ | -4 |
|----|----|---|----|
| Co | ns | е | 11 |

By signing this document, you are agreeing to be in the study. We will give you a copy of this document for your records. We will keep one copy with the study records. Be sure that we have answered any questions you have about the study and you understand what you are asked to do. You may contact the researcher or the study staff if you think of a question later.

| I agree to participate in the st | ıdy. |
|---|---|
| Printed Name | |
| Signature | Date |
| | port to teacher and/or educational team sport of my learning and memory data with my teacher |
| YES NO | |
| Signature | |
| Consent to be contacted for F I agree to be contacted for pa | articipation in Future Research ticipation in future research. |
| YES NO | |
| Signature | |